CLINICAL TRIAL: NCT06170476
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Dose-Finding Study of HSK21542 Injection for the Prevention of Postoperative Nausea and Vomiting (PONV)
Brief Title: A Clinical Trial Evaluating the Efficacy and Safety of HSK21542 in PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Mengchang Yang, Deputy Chief Physician, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSK21542-IIT-01
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HSK21542-60μg (Experimental)
  Interventions: Drug: HSK21542-60μg
- HSK21542-120μg (Experimental)
  Interventions: Drug: HSK21542-120μg
- HSK21542-180μg (Experimental)
  Interventions: Drug: HSK21542-180μg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK21542-60μg — HSK21542 injection of 60 μg was administered once within 15 min before the end of surgery, and was administered by intravenous bolus injection for no less than 30 s;
  Arms: HSK21542-60μg
Drug: HSK21542-120μg — HSK21542 injection of 120 μg was administered once within 15 min before the end of surgery, and was administered by intravenous bolus injection for no less than 30 s;
  Arms: HSK21542-120μg
Drug: HSK21542-180μg — HSK21542 injection of 180 μg was administered once within 15 min before the end of surgery, and was administered by intravenous bolus injection for no less than 30 s;
  Arms: HSK21542-180μg
Drug: Placebo — A placebo was administered once within 15 min before the end of surgery, and was administered by intravenous bolus injection for no less than 30 s;
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Dose-Finding study. About 200 subjects undergoing elective laparoscopic abdominal or gynecological surgery are planned to be enrolled and randomized into four groups by a ratio of 1:1:1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years old, male or female;
2. The American Society of Anesthesiologists (ASA) Class I-III;
3. 18 kg/m2 ≤ BMI ≤ 40 kg/m2;
4. Hospitalized subjects scheduled to undergo elective laparoscopic abdominal or gynecological surgery under general anesthesia for an expected anesthetic time of ≥ 1 h;
5. Subjects with intermediate or high risk (score ≥ 2 points) experiencing PONV judged by the investigator using the Apfel simplified risk score;
6. Subjects who agree to participate in the trial and voluntarily sign the Informed Consent Form (ICF);

Exclusion Criteria:

Prior and concomitant diseases

1. History or evidence of any of the following diseases prior to screening:

   1. Respiratory diseases: severe chronic obstructive pulmonary disease, acute exacerbation of chronic obstructive pulmonary disease, severe airway stenosis, large pharyngolaryngeal mass, (broncho) tracheoesophageal fistula or airway tear, and serious respiratory tract infection within 2 weeks prior to screening;
   2. Central nervous system disorders: subjects with epilepsy, Parkinson's disease, or other central nervous system diseases causing nausea and vomiting, such as craniocerebral injury, intracranial space-occupying lesions, intracranial aneurysms, etc.;
   3. Cardiovascular diseases: subjects with uncontrolled hypertension [systolic blood pressure (SBP) ≥170 mmHg and/or diastolic blood pressure (DBP) ≥105 mmHg without treatment with antihypertensive medication, or SBP ≥160 mmHg and/or DBP ≥100 mmHg after treatment with antihypertensive medications], serious cardiac insufficiency ( the New York Heart Association [NYHA] Grade III-IV), unstable angina pectoris, acute myocardial infarction, severe arrhythmia, history of tachycardia/bradycardia requiring medical treatment, Grade II-III atrioventricular block (excluding pacemaker use) within 6 months prior to screenin;
   4. Digestive disorders: subjects with intestinal obstruction or other digestive diseases that may cause nausea and vomiting as judged by the investigator;
   5. Patients with a confirmed diagnosis of vestibular function disorder, excluding travel sickness (including but not limited to peripheral vestibular syndrome, central vestibular syndrome, etc.);
   6. Subjects with a history of significant and chronic dizziness.

   Prior and concomitant medications
2. Any of the following medications or treatments have been used at screening:

   1. Subjects who have received antiemetics/medications with antiemetic effects within 24 h before the start of surgery or who have used antiemetics/drugs with antiemetic effects before the start of surgery for no more than 5 half-lives (calculated as the longest time);
   2. Subjects with neoplasm malignant treated with chemotherapy within 4 weeks prior to screening;

   Laboratory and other tests
3. Laboratory test indicators at screening meet the following criteria:

   1. White blood cell count < 3.0 × 109/L;
   2. Platelet count < 80 × 109/L;
   3. Hemoglobin< 70 g/L;
   4. Prolongation of prothrombin time (PT) exceeding the upper limit of normal for 3 seconds;
   5. Prolongation of activated partial thromboplastin time (APTT) exceeding the upper limit of normal for 10 seconds;
   6. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3 × ULN;
   7. Total bilirubin > 2 × ULN;
   8. Blood creatinine > 2 × ULN;
   9. Fasting serum glucose≥ 11.1 mmol/L;

   Other conditions
4. Subjects anticipated to require continued endotracheal intubation after the end of surgery;
5. Subjects anticipated to require the insertion of nasal or oral gastric tubes after the end of surgery;
6. Subjects with a history of serious drug allergies or those allergic to the investigational drugs specified in the protocol;
7. Subjects with a history of drug abuse, drug addiction, or alcoholism within 3 months prior to screening, where alcoholism is defined as consuming > 2 units of alcohol on average daily (1 unit = 360 mL of beer with 5% alcohol, 45 mL of liquor with 40% alcohol or 150 mL of wine);
8. Subjects with nausea, retching, or vomiting within 24 h prior to induction of anesthesia (except for those caused by bowel preparation);
9. Subjects who have participated in any investigational trial (defined as receiving investigational drug or placebo) within 3 months prior to screening;
10. Female subjects who are pregnant or breastfeeding; female or male subjects of child-bearing potential are unwilling to use contraception throughout the entire study period and for 3 months after the study completion;
11. Subjects judged by the investigator to be unsuitable for participating in this clinical trial for any other factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Complete response | 24 hours after the end of surgery
  The primary efficacy analysis was the complete response (CR)within the 24 hours after the end of surgery (CR was defined as no vomiting or retching and on use of rescue medication)

SECONDARY OUTCOMES:
Proportion of subjects experiencing nausea within 24 hours after the end of surgery | 24 hours after the end of surgery
  Nausea (defined as a feeling of urgency to vomit, characterized by merycism and/or urgent vomiting) measured on a 0-10 verbal response scale[VAS], where 0=no nausea at all and 10=the worst nausea that cannot be tolerated
Proportion of subjects experiencing significant nausea within 24 hours after the end of surgery | 24 hours after the end of surgery
  Significant nausea is defined as VAS score ≥ 4 cm
Proportion of subjects experiencing vomiting within 24 hours after the end of surgery | 24 hours after the end of surgery
  vomiting [even with the expulsion of scanty gastric contents] or retching [presence of vomiting muscle movement without the expulsion of gastric contents])
Proportion of subjects using rescue medication within 24 hours after the end of surgery | 24 hours after the end of surgery
  Any drug given in the post-operative period with the intention of providing anti-emetic rescue is counted as rescue anti-emetic medication
Time to first occurrence of vomiting or rescue therapy (whichever occurs first) within 24 hours after the end of surger | 24 hours after the end of surgery
  Vomiting includes vomiting or retching
The cumulative morphine doses administered within 24 hours after the end of surgery | 24 hours after the end of surgery
  Morphine as the postoperative analgesics
PONV Satisfaction Score by Subject and Investigator | 24 hours after the end of surgery
  Satisfaction Score rating range 0-10,where 0=not satisfactory at all, and 10=the most satisfactory

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Sichuan, China